CLINICAL TRIAL: NCT01381224
Title: Do Lumbar Spine Injections Improve Short-Term Biomechanical Outcomes in Patients With Chronic Low Back Pain
Brief Title: Do Lower Spine Injections Improve Outcomes for Lower Back Pain Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 629-2010
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Low Back Pain
Keywords: low back pain; lumbar; injection; lumbar pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation of biomechanical effects post injection: Observation of effects on gait, lumbar spine range of motion and pain symptoms immediately following injection and at two weeks post injection.
  Interventions: Other: Observation of biomechanical effects post injection

INTERVENTIONS:
Other: Observation of biomechanical effects post injection — Observation of effects on gait, lumbar spine range of motion and pain symptoms immediately following injection and at two weeks post injection

SUMMARY:
The purpose of this project is to determine the effect of lower back injections on select biomechanical outcomes, walking patterns, lower back flexibility and balance.

DETAILED DESCRIPTION:
The purpose of this project is to determine the effect of lumbar injections on select biomechanics parameters; walking pattern, lumbar flexibility and balance. The surveys will help assess the patient's sense of functional ability and feeling of wellness compared with low back pain scores. The long terms goals of this project will be to elucidate the mechanism of action of injections and to improve identification of patients that are likely to benefit from injection therapy

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of lumbar spine stenosis
* receiving lumbar epidural injection
* age 18-90 years
* BMI <35kg/m2
* walking unaided

Exclusion Criteria:

* age <18 or >90 years
* BMI >35 kg/m2
* severely impaired intellectual capacity
* medications that could impact balance
* dementia, or other neurodegenerative diseases that would preclude appropriate cognitive or physical ability to perform study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving a lumbar epidural steroid injection for lumbar spine stenosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Determine the immediate biomechanical effect in patients that receive a lumbar epidural injection | Immediately following injection
  We hypothesize that patients will demonstrate increased gait velocity, increased step length, decreased asymmetry and increased lumbar ROM immediately after injection compared to pre-injection

SECONDARY OUTCOMES:
Determine the short-term biomechanical effect in patients that receive a lumbar epidural injection | Two weeks following injection
  We hypothesize that patients will demonstrate increased gait velocity, increased step length, decreased asymmetry and increased lumbar ROM 2 weeks after injection compared with pre- and post-injection time points
Determine the relationship between biomechanical status before injection and short-term pain reduction | Two weeks following injection
  We hypothesize that those patients with moderate biomechanical limitation before injection (e.g., higher gait velocity, higher step length, lower asymmetry, and greater lumbar ROM) will have greater positive biomechanical response than patients who demonstrate severe biomechanical limitation pre-injection. This response to the injection will be measured by the changes in gait and lumbar spine range of motion and pain symptoms with these activities at 2 weeks after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P Conrad, Ph.D., Principal Investigator — UF Department of Orthopaedics and Rehabilitation; D J Kennedy, M.D., Principal Investigator — UF Department of Orthopaedics and Rehabilitation; Heather K Vincent, Ph.D., Principal Investigator — UF Department of Orthopaedics and Rehabilitation; Deepa Sunkari, M.D., Principal Investigator — UF Department of Orthopaedics and Rehabilitation; Amanda N Seay, B.S., Principal Investigator — UF Department of Orthopaedics and Rehabilitation
Locations (2):
- United States (2):
  - Shands Rehabilitation Hospital, Gainesville, Florida
  - UF&Shands Orthopaedics and Sports Medicine Institute, Gainesville, Florida